CLINICAL TRIAL: NCT06975072
Title: Pharmacokinetics and Impact of Magnesium Sulfate on Neuromonitoring in Spinal Surgery
Brief Title: Effect of Magnesium on Neuromonitoring
Acronym: MgNm
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 25-43430
Record Dates: First submitted 2025-03-31; First posted 2025-05-16 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Spine; Pain; Spine Surgery; Spine Surgery With Neuromonitoring; Spine Surgery With Motor Evoked Potential Monitoring; Spine Fusion
Keywords: spine; spine surgery; spine fusion; magnesium; neuromonitoring; motor evoked potential monitoring
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Magnesium Arm (Experimental): A single intravenous bolus of Mg of 30mg/kg (based on ideal body weight) will be administered over a period of 10 minutes (min).
  Interventions: Drug: Magnesium sulfate administration

INTERVENTIONS:
Drug: Magnesium sulfate administration — A single intravenous bolus of Mg of 30mg/kg (based on ideal body weight) will be administered over a period of 10 minutes (min).

SUMMARY:
Intraoperative neurophysiologic monitoring (IONM) is commonly used during complex spinal surgery to monitor the integrity of neural structures and improve the perioperative safety profile. Transcranial Motor Evoked Potentials (TcMEPs) monitor the integrity of the motor pathways and are one of the most commonly used monitoring modalities in spinal surgery. Because inhaled anesthetics can negatively affect the ability to monitor TcMEPs, anesthesiologists commonly use a combination of propofol and opioids to maintain the anesthetic state. Additionally, anesthesiologists will frequently administer intravenous infusions of medications that can decrease postoperative pain and opioid use (called opioid-sparing adjuncts) because spinal surgeries result in significant postoperative pain. Despite the increasing use of these agents, there is scant clinical data about how they may affect the integrity of TcMEP monitoring. Magnesium (Mg), a N-methyl-d-aspartate receptors (NMDA) receptor antagonist, is one of the adjuncts with robust data supporting clinical efficacy to decrease pain and opioid use on TcMEPs. Mg has been used clinically for decades. The investigators commonly utilize intravenous magnesium as a component of our spinal anesthesia protocol. However, there is only a single case report that discusses the effects of Mg on TcMEPs. Here the investigators propose a prospective clinical trial to quantitatively assess the effects of various Mg plasma levels on TcMEPs. There is a lack of literature on the pharmacokinetics of magnesium in non-pregnant patients.

DETAILED DESCRIPTION:
Spinal surgeries continue to increase in frequency and complexity, with the potential to cause injury to neural structures. Intraoperative neurophysiologic monitoring (IONM) is a crucial tool in spinal surgery, offering real-time detection of adverse changes in the integrity of neural systems governing sensory and motor function. At the same time, the patient is anesthetized, which decreases the risk of permanent and severe neuronal injury. Transcranial Motor Evoked Potentials (TcMEPs), which involve nonspecific stimulation of pyramidal axons in the cerebral motor cortex while monitoring myogenic responses in various muscle groups, are the most common IONM technique during complex spinal surgeries to assess the integrity of motor pathways. Injury to either the cord or nerve roots is detected as a change in the amplitude or latency of the myogenic response, and this test has very high sensitivity and specificity for injury. Many factors, such as hypotension, hypothermia, anemia, and anesthetics, can affect the amplitude/ latency of TcMEPs. Early during the development of this monitoring modality, it was recognized that volatile inhaled anesthetics severely inhibited the ability to elicit reliable TcMEP data. Clinical trials showed that using propofol, an intravenous (iv) general anesthetic, combined with moderate doses of opioids facilitated high-quality IONM while providing appropriate anesthetic conditions for surgery. While the propofol/opioid combination became the "default" anesthetic as the frequency of IONM increased, there was increasing recognition that anesthesiologists could enhance the perioperative recovery profile by adding iv opioid-sparing adjuncts like ketamine, lidocaine, and magnesium (Mg) to the intraoperative regimen. Furthermore, with the development of enhanced recovery after surgery (ERAS) protocols, nearly all spinal surgeries (except for the most minor procedures) now utilize at least one of these adjuncts. However, while these agents are increasingly used for spinal surgeries, there is scant clinical data about how they may affect the integrity of TcMEP monitoring. High-quality IONM monitoring is invaluable for improving the perioperative safety profile of patients undergoing spinal surgery. However, there is a lack of rigorous quantitative data on the effects of anesthetic adjuncts on TcMEPs. Therefore, the investigators seek to establish a robust protocol that can be used quantitively to determine the impact of these agents on TcMEPs. Our overall hypothesis is that anesthetic adjuncts can variably affect TcMEPs. To establish this protocol, the investigators selected Mg to develop and optimize our protocol. Mg, an NMDA receptor antagonist, is commonly used to reduce postoperative pain and opioid use during major spinal surgery; however, to date, there is only a single case report that discusses the effects of Mg on TcMEPs. However, substantial literature shows that Mg can adversely affect neuromuscular physiology, including through decreased release of acetylcholine from presynaptic neurons and by directly suppressing current flux through muscle-based nicotinic acetylcholine receptors. These effects may explain the clinical observation that higher Mg doses can dose-dependently suppress TcMEPs. While there is a similar dearth of information regarding the effect of the other anesthetic adjuncts on TcMEPs, the investigators propose to begin our investigation and protocol optimization with Mg because of its long use in clinical practice, its safety profile, its effectiveness as an opioid-sparing adjunct, the frequency with which it is used in spinal surgery (an estimated frequency of >75% of patients that receive IONM and the dearth of quantitative data on its effects on TcMEPs. The optimized protocol and initial data will support a more extensive future trial to systemically characterize the effects of all the common anesthetic adjuncts on TcMEPs. High-quality data that quantitatively determine the effects of Mg on TcMEPs will allow clinicians to rationally select effective doses that provide analgesia while ensuring high-quality intraoperative monitoring.

Patient Recruitment: The investigators will use the surgical schedule and CaseView to screen for eligible patients. The PI will determine eligibility by a medical record review, performed prior to the patients surgery and attempts at patient contact. Eligibility will be determined according to the criteria listed in the relevant sections. Briefly, eligible patients are adults >18 years of age, presenting for elective spinal fusion procedures. Before the investigators begin recruitment, all surgeons involved with spine surgery will be contacted by email to inform them about the study and to receive approval for their patients to participate. After each patient has provided informed consent, the investigators will contact the surgeons by email to inform them of the patient's participation.

Consent: The investigators will attempt to obtain eConsent from study subjects prior to arrival at the hospital, however, this may not be possible in all situations. Some of our patients may consent to the procedure, but be unable to complete the eConsent process prior to arrival because of a lack of technical capacity. Day of surgery written consent will only be used as a last resort if the investigators are unable to obtain eConsent. The investigators will obtain verbal consent at least 1 day prior to the scheduled procedure for any patient that cannot provide eConsent, and then obtain written hard copy consent on the day of surgery.

Operating Room: All study patients will undergo general anesthesia like non-study patients. The anesthesia time will not be extended for any study-related activities. The investigators will complete study-related activities during the anesthesia and surgery time without interrupting the standard care.

All patients will receive a standardized anesthetic, an intravenous anesthetic consisting of only propofol (60-150 mcg/kg/min) and remifentanil (0.1-0.3mcg/kg/min. Propofol will be titrated to achieve a Patient State Index (PSI) between 25 and 50 as measured using a standard SEDline Brain Function Monitor (Masimo, Inc., Irvine, CA). Anesthesiologists will be asked to avoid electroencephalographic burst suppression by adjusting the dose of propofol since prior studies have shown that burst suppression can interfere with TcMEPs. This is a standard anesthesia care for our patient care protocol and the investigators would like to avoid electroencephalographic burst suppression in patients undergoing general anesthesia. Patient will have the necessary equipment for neuromonitoring placed. These pieces of equipment are placed identically for patients who are or are not in our study, and the investigators will not add any additional monitors. All patients participating in the study will have neuromonitoring as part of their surgery, so this is not an additional study-specific procedure. Baseline motor-evoked potential data will then be collected. This baseline data is also standard practice and not a study-specific procedure. After the baseline data is collected, the investigators will commence with the study protocol. A single intravenous bolus of Mg of 30mg/kg (based on ideal body weight) will be administered over a period of 10 minutes (min).

Mg plasma levels: Blood samples will be collected to measure plasma magnesium (Mg) levels at the following time points: 0 min (pre-Mg administration), 1 min, 10 min (end of infusion), 20 min, 30 min, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, and 12 hr. The dosing and blood sampling intervals were determined by the reported half-life of Mg and in consultation with our pharmacology consultant. Blood will be sent to the UCSF Clinical laboratory.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (>18 years of age) undergoing open thoracolumbar fusion with planned neuromonitoring

Exclusion Criteria:

1. Patients with a history of significant cardiac disease (LVEF <35%, 2nd/3rd-degree block without a pacemaker, or significant arrhythmia)
2. Patients with kidney disease (GFR <30), or hepatic dysfunction (history of cirrhosis)
3. Allergy or sensitivity to magnesium
4. Patient with neuromuscular disease such as myasthenia graves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Serum Magnesium level | Through study completion, an average of 1 year
  Serum magnesium level will be measured by UCSF Lab.
Magnesium- Pharmakokinetics Clearance (CL) | Through study completion, an average of 1 year
  Serum magnesium level will be measured by UCSF Lab. Then the investigators will run the Pharmakokinetics clearance (CL) data with the levels.
Magnesium- Pharmacokinetics central volume of distribution (Vc) | Through study completion, an average of 1 year
  Serum magnesium level will be measured by UCSF Lab. Then the investigators will run the Pharmacokinetics Central volume of distribution (Vc) data with the levels.
Magnesium- Pharmakokinetics (PK) intercompartmental clearance (Q) | Through study completion, an average of 1 year
  Serum magnesium level will be measured by UCSF Lab. Then the investigators will run the PK intercompartmental clearance (Q) data with the levels.
Magnesium- Pharmakokinetics peripheral volume of distribution (Vp) | Through study completion, an average of 1 year
  Serum magnesium level will be measured by UCSF Lab. Then the investigators will run the PK peripheral volume of distribution (Vp) data with the levels.

SECONDARY OUTCOMES:
Neuromonitoring data-Stimulation voltage | Through study completion, an average of 1 year
  The investigators will change in stimulation voltage in different time points using the students t-test
Neuromonitoring data- motor-evoked potential (MEP) amplitude | Through study completion, an average of 1 year
  The investigators will compare motor-evoked potential (MEP) amplitude responses at different time points using the students t-test.
Neuromonitoring data- Motor Evoked Potential (MEP) Latency | Through study completion, an average of 1 year
  The investigators will compare the change in MEP latency using the students t-test

CONTACTS AND LOCATIONS:
Overall Officials: Hemra Cil, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Blacker SN, Vincent A, Burbridge M, Bustillo M, Hazard SW, Heller BJ, Nadler JW, Sullo E, Lele AV; Society for Neuroscience in Anesthesiology and Critical Care. Perioperative Care of Patients Undergoing Major Complex Spinal Instrumentation Surgery: Clinical Practice Guidelines From the Society for Neuroscience in Anesthesiology and Critical Care. J Neurosurg Anesthesiol. 2022 Jul 1;34(3):257-276. doi: 10.1097/ANA.0000000000000799. Epub 2021 Sep 6. PMID 34483301
- [Background] Johnson T, Kale EB, Husain AM. Magnesium Sulfate-Induced Motor Evoked Potential Changes. Neurodiagn J. 2018;58(2):83-90. doi: 10.1080/21646821.2018.1469336. PMID 29923809
- [Background] Wang H, Liang QS, Cheng LR, Li XH, Fu W, Dai WT, Li ST. Magnesium sulfate enhances non-depolarizing muscle relaxant vecuronium action at adult muscle-type nicotinic acetylcholine receptor in vitro. Acta Pharmacol Sin. 2011 Dec;32(12):1454-9. doi: 10.1038/aps.2011.117. Epub 2011 Oct 10. PMID 21986576
- [Background] Yue L, Lin ZM, Mu GZ, Sun HL. Impact of intraoperative intravenous magnesium on spine surgery: A systematic review and meta-analysis of randomized controlled trials. EClinicalMedicine. 2022 Jan 5;43:101246. doi: 10.1016/j.eclinm.2021.101246. eCollection 2022 Jan. PMID 35028543
- [Background] Martell BA, Arnsten JH, Krantz MJ, Gourevitch MN. Impact of methadone treatment on cardiac repolarization and conduction in opioid users. Am J Cardiol. 2005 Apr 1;95(7):915-8. doi: 10.1016/j.amjcard.2004.11.055. PMID 15781034
- [Background] Furutani K, Deguchi H, Matsuhashi M, Mitsuma Y, Kamiya Y, Baba H. A Bolus Dose of Ketamine Reduces the Amplitude of the Transcranial Electrical Motor-evoked Potential: A Randomized, Double-blinded, Placebo-controlled Study. J Neurosurg Anesthesiol. 2021 Jul 1;33(3):230-238. doi: 10.1097/ANA.0000000000000653. PMID 31633576
- [Background] Tramer MR, Schneider J, Marti RA, Rifat K. Role of magnesium sulfate in postoperative analgesia. Anesthesiology. 1996 Feb;84(2):340-7. doi: 10.1097/00000542-199602000-00011. PMID 8602664
- [Background] Herdmann J, Deletis V, Edmonds HL Jr, Morota N. Spinal cord and nerve root monitoring in spine surgery and related procedures. Spine (Phila Pa 1976). 1996 Apr 1;21(7):879-85. doi: 10.1097/00007632-199604010-00023. PMID 8779023
- [Background] Sloan TB, Heyer EJ. Anesthesia for intraoperative neurophysiologic monitoring of the spinal cord. J Clin Neurophysiol. 2002 Oct;19(5):430-43. doi: 10.1097/00004691-200210000-00006. PMID 12477988
- [Background] Macdonald DB, Skinner S, Shils J, Yingling C; American Society of Neurophysiological Monitoring. Intraoperative motor evoked potential monitoring - a position statement by the American Society of Neurophysiological Monitoring. Clin Neurophysiol. 2013 Dec;124(12):2291-316. doi: 10.1016/j.clinph.2013.07.025. Epub 2013 Sep 18. PMID 24055297